CLINICAL TRIAL: NCT02663622
Title: A Phase II Trial of CD24Fc for Prevention of Acute Graft-versus-Host Disease Following Myeloablative Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Phase II Trial of Efprezimod Alfa (CD24Fc, MK-7110) for the Prevention of Acute Graft-Versus-Host Disease (GVHD) Following Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) (MK-7110-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncoimmune, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Ohio State University (Other); University of Michigan Rogel Cancer Center (Other); Indiana University School of Medicine (Other); Barbara Ann Karmanos Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7110-002; HUM00107805 (Other: University of Michigan); 15-4789 (Other: Orphan Drug Designation); R44CA221513 (NIH); R44CA246991 (NIH); UMCC 2015.181 (Other: UMCC); MK-7110-002 (Other: Merck Protocol Number); NCI-2017-00017 (Other: National Cancer Institute); CD24Fc-002 (Other: OncoImmune Protocol Number)
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Graft Versus Host Disease; Hematopoietic Stem Cell Transplantation; Leukemia
MeSH Terms: conditions — Graft vs Host Disease; Leukemia | interventions — Methotrexate; Tacrolimus; Saline Solution

STUDY DESIGN:
Intervention Model Description: Study was double blind for the first 6 participants in each arm. At that point, the recommended phase II dose (RP2D) was determined, and the selected arm enrolled additional participants in an open label fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Efprezimod alfa 240 mg (Experimental): Efprezimod alfa in 240 mg as intravenous (IV) infusion at Day -1 + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
  Interventions: Drug: Efprezimod alfa; Drug: Methotrexate; Drug: Tacrolimus
- Efprezimod alfa 480 mg (Experimental): Efprezimod alfa in 480 mg as intravenous (IV) infusion at Day -1 + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
  Interventions: Drug: Efprezimod alfa; Drug: Methotrexate; Drug: Tacrolimus
- Efprezimod alfa 960 mg (Experimental): Efprezimod alfa (480 mg (day -1), 240 mg (day +14) and 240 mg (day +28)) + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
  Interventions: Drug: Efprezimod alfa; Drug: Methotrexate; Drug: Tacrolimus
- Placebo (Placebo Comparator): Placebo to efprezimod alfa (saline IV injection solution) on day -1 or days -1, 14, and 28 + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
  Interventions: Drug: Methotrexate; Drug: Tacrolimus; Drug: Placebo

INTERVENTIONS:
Drug: Efprezimod alfa — Acute GVHD prophylaxis
  Other Names: CD24 Fusion Protein; MK-7110
  Arms: Efprezimod alfa 240 mg; Efprezimod alfa 480 mg; Efprezimod alfa 960 mg
Drug: Methotrexate — Acute GVHD prophylaxis
  Other Names: Trexall
Drug: Tacrolimus — Acute GVHD prophylaxis
  Other Names: FK506; Prograf
Drug: Placebo — 100 ml saline IV infusion.
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
This is a multicenter prospective phase IIa dose escalation and phase IIa expansion cohort clinical trial designed to evaluate the safety and tolerability of efprezimod alfa for acute GVHD prophylaxis.

DETAILED DESCRIPTION:
The first part of this study was a phase IIa randomized, double blind, placebo controlled, multi-center study to investigate adding efprezimod alfa to standard of care tacrolimus and methotrexate in acute graft-versus host disease (GVHD) prophylaxis for allogeneic hematopoietic stem cell transplantation (HCT) with matched unrelated donors in treatment of leukemia and myelodysplastic syndrome. The primary objective was to evaluate the safety, tolerability and dose-limiting toxicities (DLTs) of efprezimod alfa in participants undergoing matched unrelated donor myeloablative allogeneic HCT for malignant hematologic disorders. Three dose cohorts were planned with 240 mg at day -1 (one day prior to HCT), 480 mg at day -1, and the multi-dose cohort of 480-240-240 mg at day -1, day 14 and day 28. The efprezimod alfa : placebo randomization ratio was 3:1.

The second part was a prospective open label phase IIa expansion cohort trial investigating the addition of efprezimod alfa to standard acute graft-versus host disease (GVHD) prophylaxis for allogeneic hematopoietic stem cell transplantation (HCT). Based on the first part's safety results and the pharmacokinetic data, the phase IIa expansion dose was the multi-dose 480-240-240 mg regimen administered on day -1, day 14 and day 28, respectively. The primary objective of phase IIa expansion was to determine if the addition of efprezimod alfa to standard GVHD prophylaxis improves 180 days post-HCT grade III-IV acute GVHD-free survival (AGFS) when compared to Center for International Blood and Marrow Transplant Research (CIBMTR) database registered control participants who had standard GVHD prophylaxis alone. Eligible participants were those requiring allogeneic HCT for malignant hematologic conditions and receiving a myeloablative conditioning regimen.

ELIGIBILITY:
Inclusion Criteria

4.1.1 A prospective participant for allogeneic hematopoietic stem cell transplantation (HCT) for a malignant hematologic disorder.

4.1.2 The donor and recipient must have a human leukocyte antigen (HLA)-8/8 allelic match at the HLA-A, -B, -C, and - DRB1 loci. High-resolution typing is required for all alleles for unmatched donors. Only matched unrelated donors are acceptable for this trial.

4.1.3 The following diagnoses are to be included:

1. Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) in first or second remission. Remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment, < 5% blasts in the bone marrow and absence of extramedullary disease including central nervous system (CNS) involvement.
2. Chronic Myelogenous Leukemia (CML) in first or subsequent chronic phase failing to respond (or intolerant) to at least two different tyrosine kinase inhibitors. CML in accelerated or blast phase (CML-AP/BP) are eligible without requirement to fail tyrosine kinase inhibitor therapy, but must be in remission at time of enrollment. Remission is defined as the absence of blasts in the peripheral circulation at the time of enrollment, < 5% blasts in the bone marrow and absence of extramedullary disease including CNS involvement.
3. Myelodysplastic syndrome (MDS) with intermediate or high-risk International Prognostic Scoring System (IPSS) or equivalent Revised IPSS (IPSS-R) score with < 10% blasts in the bone marrow.
4. Chronic Myelomonocytic Leukemia (CMML) with < 10% blasts in the bone marrow.

4.1.4 Males or non-pregnant, non-lactating females, ≥ 18 years of age. Note there is no defined upper age limited, so long as deemed appropriate candidate for myeloablative conditioning.

4.1.5 Karnofsky Performance Status >70%.

4.1.6 Participants must have normal or near normal organ function as defined by their treating institutions bone marrow transplantation (BMT) program clinical practice guidelines. In addition, for purposes of this protocol minimum organ function criteria within 21 days of beginning conditioning include:

TABLE 1: Eligibility According to Pre HCT Organ Function Total bilirubin ≤2.5 mg% (unless from Gilbert's disease or disease-related) Aspartate aminotransferase (serum glutamic-oxaloacetic transaminase) (AST[SGOT])/ alanine aminotransferase (serum glutamic-pyruvic transaminase) (ALT[SGPT]) <3.0 X institutional upper limit of normal Estimated or actual glomerular filtration rate (GFR) >50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal (GFR should be corrected for body surface area [BSA]) Pulmonary Function Tests* diffusing capacity of the lung for carbon monoxide (DLCO), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) > 50% DLCO should be corrected for hemoglobin Ejection Fraction* >50% Hematopoietic Cell Transplantation-Specific Comorbidity Index (HCT-CI) ≤ 5

*May be assessed up to 6 weeks prior to the start of conditioning therapy

4.1.7 Ability to understand and the willingness to sign a written informed consent document.

4.1.8 Women of child bearing potential and men must agree to use contraception prior to study entry and through day 100 post HCT (hormonal or barrier method of birth control; abstinence). Should a woman become pregnant or suspect she is pregnant while she or her partner is on treatment in this study, she should inform her study physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study until day 100 post HCT.

Exclusion Criteria:

4.2.1 Participants may not have presence of active CNS disease or extramedullary disease.

4.2.2 Prior cytotoxic chemotherapy within 21 days from the initiation of HCT conditioning (i.e. intensive induction / consolidation for AML). Note, certain low intensity treatments not intended to induce remission but rather stabilize disease are acceptable up to 24 hrs prior to initiation of HCT conditioning (i.e. Tyrosine Kinase Inhibitor, sorafenib).

4.2.3 Cord blood and haploidentical donors are not eligible.

4.2.4 HLA-mismatch at the HLA-A, -B, -C, and - DRB1 loci. Note, HLA-DQ mismatches are permissible.

4.2.5 Pregnant and nursing mothers are excluded from this study. This is because the risk to the fetus is unknown.

4.2.6 Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the participant or raise concern that the participant would not comply with protocol procedures.

4.2.7 Uncontrolled infections. Participants still under therapy for presumed or proven infection are eligible provided there is clear evidence (radiologic, clinical and/or culture) that the infection is well controlled.

4.2.8 Participants seropositive or polymerase chain reaction (PCR) positive for the human immunodeficiency virus (HIV). Participants with evidence of Hepatitis B or Hepatitis C PCR positivity.

4.2.9 Prior HCT (allograft or prior autograft).

4.2.10 Use of T cell depletion either ex vivo or in vivo (i.e. anti-thymocyte globulin [ATG], alemtuzumab) is prohibited.

4.2.11 Current or prior diagnosis of antecedent Myelofibrosis is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Toubai T, Rossi C, Oravecz-Wilson K, Zajac C, Liu C, Braun T, Fujiwara H, Wu J, Sun Y, Brabbs S, Tamaki H, Magenau J, Zheng P, Liu Y, Reddy P. Siglec-G represses DAMP-mediated effects on T cells. JCI Insight. 2017 Jul 20;2(14):e92293. doi: 10.1172/jci.insight.92293. eCollection 2017 Jul 20. PMID 28724800
- [Background] Toubai T, Hou G, Mathewson N, Liu C, Wang Y, Oravecz-Wilson K, Cummings E, Rossi C, Evers R, Sun Y, Wu J, Choi SW, Fang D, Zheng P, Liu Y, Reddy P. Siglec-G-CD24 axis controls the severity of graft-versus-host disease in mice. Blood. 2014 May 29;123(22):3512-23. doi: 10.1182/blood-2013-12-545335. Epub 2014 Apr 2. PMID 24695850
- [Background] Toubai T, Mathewson ND, Magenau J, Reddy P. Danger Signals and Graft-versus-host Disease: Current Understanding and Future Perspectives. Front Immunol. 2016 Nov 29;7:539. doi: 10.3389/fimmu.2016.00539. eCollection 2016. PMID 27965667
- [Result] Magenau J, Jaglowski S, Uberti J, Farag SS, Riwes MM, Pawarode A, Anand S, Ghosh M, Maciejewski J, Braun T, Devenport M, Lu S, Banerjee B, DaSilva C, Devine S, Zhang MJ, Burns LJ, Liu Y, Zheng P, Reddy P. A phase 2 trial of CD24Fc for prevention of graft-versus-host disease. Blood. 2024 Jan 4;143(1):21-31. doi: 10.1182/blood.2023020250. PMID 37647633
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The CD24Fc 960 mg arm was initiated alongside the other 3 arms. Once the recommended phase 2 dose (RP2D) was determined, the other 3 arms ceased recruitment but additional participants were recruited into the CD24Fc 960 mg arm. Per FDA request, all participants in the CD24Fc 960 mg arm are considered a single population.
Groups:
- Placebo: Placebo to CD24Fc (saline IV injection solution) on day -1 or days -1, 14, and 28 + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
- CD24Fc 240 mg: CD24Fc in 240 mg as intravenous (IV) infusion at Day -1 + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
- CD24Fc 480 mg: CD24Fc in 480 mg as intravenous (IV) infusion at Day -1 + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
- CD24Fc 960 mg: CD24Fc (480 mg (day -1), 240 mg (day +14) and 240 mg (day +28)) + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
Period: Overall Study
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Started | 6 | 6 | 6 | 26
Completed | 3 | 5 | 5 | 17
Not Completed | 3 | 1 | 1 | 9
Not completed — Death | 3 | 1 | 1 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 26 | 44
Age, Customized [Count of Participants; unit: Participants]
  18-29 years of age | 0 | 1 | 2 | 3 | 6
  30-39 years of age | 1 | 0 | 0 | 3 | 4
  40-49 years of age | 1 | 1 | 0 | 4 | 6
  50-59 years of age | 2 | 0 | 0 | 8 | 10
  ≥60 years of age | 2 | 4 | 4 | 8 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 12 | 18
  Male | 4 | 4 | 4 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 6 | 26 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 5 | 6 | 25 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE is presented. As described in the protocol, AEs reported after the protocol-specified timeframe were not analyzed in this outcome measure: 1 day prior to hematopoietic stem cell transplantation (HCT) through either 30 or 60 days post-HCT, depending on arm as defined in the Time Frame section.
Time Frame: Up to approximately 32 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms. Up to approximately 62 days for the CD24Fc 960 mg arm.
Population: All participants who enrolled prior to determination of the recommended phase II dose and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 6 | 6 | 6 | 6

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: 1 day for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms. Up to approximately 30 days for the CD24Fc 960 mg arm.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: A DLT was defined as: any Grade III or higher non-hematologic toxicity not clearly related to the underlying malignancy, intercurrent infection, or the hematopoietic stem cell transplantation conditioning regimen; any death not related to relapse or intercurrent infection; and failure to engraft by day 30. Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. Hypersensitivity reactions and other infusion-related reactions were not considered DLTs.
Time Frame: Up to 32 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms. Up to 62 days for the CD24Fc 960 mg arm.
Population: All participants who enrolled prior to determination of the recommended phase II dose, received at least one dose of study drug, and completed the protocol's DLT evaluation period were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Open Label Expansion Arm Only: Grade III-IV Acute Graft-Versus-Host Disease (GVHD) Free Survival (AGFS)
Description: AGFS was defined as the time from the date of hematopoietic stem cell transplantation (HCT) to the earliest of Grade III-IV acute GVHD or death due to any cause, whichever occurred first. Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. Participants were censored at 181 days.
Time Frame: Up to 181 days
Population: Per protocol, only participants enrolled in the CD24Fc 960 mg arm (from both the dose escalation and expansion phases) who received at least one dose of study drug and underwent HCT were analyzed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CD24Fc 960 mg
Number analyzed (Participants) | 26
Days | 159.0 (46.86)
Statistical Analysis 1: Comparison: CD24Fc 960 mg; A hazard ratio was calculated based on a Cox proportional hazards regression model with treatment as a factor using the robust sandwich covariance estimator, comparing the CD24Fc 960 mg arm to a matched control group consisting of 92 participants from the Center for International Blood and Marrow Transplant Research (CIBMTR) observational databases of clinical information on HCT, whose mean grade III-IV AGFS in days was 135.8 with an SD of 64.66; Test type: Superiority; p = 0.0274, Log Rank; Log-rank test stratified by the matched sets; Cox Proportional Hazard = 0.13, 95% CI 2-sided [0.01 to 0.62]

5. Secondary Outcome: Grade II-IV Acute Graft-Versus-Host Disease (GVHD) Free Survival (AGFS)
Description: AGFS was defined as the time from the date of hematopoietic stem cell transplantation (HCT) to the earliest of Grade II-IV acute GVHD or death due to any cause, whichever occurred first. Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. Participants were censored at 195 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms, and at 181 days for the CD24Fc 960 mg arm.
Time Frame: Up to 195 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms. Up to 181 days for the CD24Fc 960 mg arm.
Population: All participants who received at least one dose of study drug and underwent HCT were analyzed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 26
Days | 144.2 (74.98) | 145.7 (77.01) | 116.2 (86.69) | 125.4 (64.93)
Statistical Analysis 1: Comparison: CD24Fc 960 mg; A hazard ratio was calculated based on a Cox proportional hazards regression model with treatment as a factor using the robust sandwich covariance estimator, comparing the CD24Fc 960 mg arm to a matched control group consisting of 92 participants from the Center for International Blood and Marrow Transplant Research (CIBMTR) observational databases of clinical information on HCT, whose mean grade II-IV AGFS in days was 104.7 with an SD of 72.28; Test type: Superiority; p = 0.0988, Log Rank; Cox Proportional Hazard = 0.57, 95% CI 2-sided [0.30 to 1.08]

6. Secondary Outcome: Percentage of Participants Experiencing Grade II to IV Acute GVHD Following HCT
Description: The percentage of participants who experienced grade II to IV acute GVHD is presented as cumulative incidence of Grade II to IV acute GVHD by approximately 108 days following HCT. Event grading was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 criteria. The cumulative incidence (%) of acute GVHD and the 95% CI were estimated using the cumulative incidence function with death without Grade II to IV acute GVHD as a competing risk.
Time Frame: Up to approximately 108 days
Population: All participants who enrolled prior to determination of the recommended phase II dose, received at least one dose of study drug, and underwent HCT were analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Participants | 16.7 [0.5 to 54.9] | 33.3 [3.2 to 70.4] | 50.0 [7.7 to 82.9] | 33.3 [3.2 to 70.4]

7. Secondary Outcome: Percentage of Participants Experiencing Chronic GVHD Following HCT
Description: The percentage of participants who experienced chronic GVHD will be presented as cumulative incidence of chronic GVHD. Chronic GVHD assessments occurred approximately quarterly beginning on Day 100 after HCT until 1 year after HCT. The cumulative incidence (%) of chronic GVHD at 1 year post-HCT and the 95% CI were estimated using the cumulative incidence function with death without chronic GVHD as a competing risk. If the maximum observed time was <Study Day 380, the cumulative incidence at the maximum observed time is presented for a treatment group.
Time Frame: Up to 380 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Participants | 33.3 [2.5 to 72.0] | 50.0 [7.0 to 83.5] | 50.0 [6.9 to 83.6] | 83.3 [0.5 to 99.4]

8. Secondary Outcome: Percentage of Participants Experiencing Relapse Following HCT
Description: The percentage of participants who experienced relapse of disease is presented as cumulative incidence of relapse. The cumulative incidence (%) of relapse at approximately 1 year following HCT and the 95% CI were estimated using the cumulative incidence function with death without relapse as a competing risk. If the maximum observed time is < Study Day 380, the cumulative incidence at the maximum observed time is presented.
Time Frame: Up to 380 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Participants | 33.3 [2.9 to 71.1] | 0.0 [NA to NA] — The upper and lower limits are not estimable because the 95% CI is obtained using the log-log transformation. Since the estimate is 0, the CI is not estimable. | 16.7 [0.5 to 54.9] | 16.7 [0.5 to 54.9]

9. Secondary Outcome: Percentage of Participants Experiencing Non-Relapse Mortality (NRM) Following HCT
Description: The percentage of participants who experienced NRM is presented as cumulative incidence of NRM. The cumulative incidence (%) of NRM at approximately 1 year following HCT and the 95% CI were estimated using the cumulative incidence function with relapse as a competing risk. If the maximum observed time is < Study Day 380, the cumulative incidence at the maximum observed time will be presented.
Time Frame: Up to 380 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Participants | 16.7 [0.5 to 54.9] | 16.7 [0.5 to 54.9] | 0.0 [NA to NA] — The upper and lower limits are not estimable because the 95% CI is obtained using the log-log transformation. Since the estimate is 0, the CI is not estimable. | 0.0 [NA to NA] — The upper and lower limits are not estimable because the 95% CI is obtained using the log-log transformation. Since the estimate is 0, the CI is not estimable.

10. Secondary Outcome: Percentage of Participants Experiencing Infection Following Hematopoietic Stem Cell Transplantation (HCT)
Description: The percentage of participants who experienced infection by approximately 101 days following HCT is presented.
Time Frame: Up to approximately 101 days
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of Participants | 33.3 | 83.3 | 33.3 | 100.0

11. Secondary Outcome: Overall Survival (OS) Following Hematopoietic Stem Cell Transplantation (HCT)
Description: OS is defined as the time from HCT to death due to any cause. Participants were censored at 380 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms, and at 366 days for the CD24Fc 960 mg arm.
Time Frame: Up to 380 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms. Up to 366 days for the CD24Fc 960 mg arm.
Population: All participants who received at least one dose of study drug and underwent HCT were analyzed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 26
Days | 276.3 (132.25) | 343.0 (64.34) | 343.5 (72.45) | 321.2 (97.62)
Statistical Analysis 1: Comparison: CD24Fc 960 mg; A hazard ratio was calculated based on a Cox proportional hazards regression model with treatment as a factor using the robust sandwich covariance estimator, comparing the CD24Fc 960 mg arm to a matched control group consisting of 92 participants from the Center for International Blood and Marrow Transplant Research (CIBMTR) observational databases of clinical information on HCT, whose mean OS in days was 319.3 with an SD of 93.83; Test type: Superiority; p = 0.9088, Log Rank; Cox Proportional Hazard = 1.12, 95% CI 2-sided [0.43 to 2.88]

12. Secondary Outcome: GVHD-Free and Relapse-Free Survival (GRFS) Following HCT
Description: This GRFS following HCT is a composite endpoint in which events included Grade III to IV acute GVHD, chronic GVHD requiring systemic immunosuppressive therapy, relapse, or death from any cause
Time Frame: Up to 380 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Days | 178.7 (151.48) | 260.5 (99.54) | 250.3 (149.68) | 227.2 (123.63)

13. Secondary Outcome: Relapse-Free Survival (RFS) Following Hematopoietic Stem Cell Transplantation (HCT)
Description: RFS is defined as the time from HCT to relapse or death due to any cause. Participants were censored at 380 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms, and at 366 days for the CD24Fc 960 mg arm.
Time Frame: Up to 380 days for the Placebo, CD24Fc 240 mg, and CD24Fc 480 mg arms. Up to 366 days for the CD24Fc 960 mg arm
Population: All participants who received at least one dose of study drug and underwent HCT were analyzed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 26
Days | 232.7 (152.48) | 342.5 (64.11) | 335.2 (92.82) | 296.2 (119.06)
Statistical Analysis 1: Comparison: CD24Fc 960 mg; A hazard ratio was calculated based on a Cox proportional hazards regression model with treatment as a factor using the robust sandwich covariance estimator, comparing the CD24Fc 960 mg arm to a matched control group consisting of 92 participants from the Center for International Blood and Marrow Transplant Research (CIBMTR) observational databases of clinical information on HCT, whose mean RFS in days was 296.0 with an SD of 115.32; Test type: Superiority; p = 0.6131, Log Rank; Cox Proportional Hazard = 1.27, 95% CI 2-sided [0.66 to 2.46]

ADVERSE EVENTS:
Time Frame: Up to 1134 days for All-Cause Mortality. Up to 1131 days for all adverse events.
Groups:
- CD24Fc 960 mg (Multi-dose): CD24Fc (480 mg (day -1), 240 mg (day +14) and 240 mg (day +28)) + Tacrolimus (begin on day -3. IV [0.03 mg/kg/day] or PO [0.045 mg/kg/dose] dosing is permitted) + Methotrexate (given intravenously at a dose of 15 mg/square meter/dose once daily on Day 1 after HCT, and at a dose of 10 mg/square meter/dose on days 3, 6, and 11 after HCT)
Arm/Group | Placebo | CD24Fc 240 mg | CD24Fc 480 mg | CD24Fc 960 mg (Multi-dose)
All-Cause Mortality (participants affected / at risk) | 3/6 | 1/6 | 1/6 | 8/26
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 1/6 | 12/26
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | CD24Fc 240 mg (N=6) | CD24Fc 480 mg (N=6) | CD24Fc 960 mg (Multi-dose) (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | CD24Fc 240 mg (N=6) | CD24Fc 480 mg (N=6) | CD24Fc 960 mg (Multi-dose) (N=26)
Anaemia (Blood and lymphatic system disorders) | 4 (15) | 6 (29) | 5 (18) | 22 (89)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 7 (9)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 2 (2) | 4 (6) | 18 (23)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (5) | 9 (9)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (19) | 6 (13) | 6 (18) | 25 (46)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3) | 9 (11)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (3) | 3 (3) | 2 (2) | 10 (11)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 11 (21)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (4) | 3 (6) | 1 (1) | 13 (31)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (7) | 1 (1) | 11 (23)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 4 (5)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 7 (8)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 3 (18) | 6 (27) | 5 (15) | 4 (10)
Neutrophil count decreased (Investigations) | 3 (11) | 5 (19) | 6 (20) | 21 (66)
Platelet count decreased (Investigations) | 5 (21) | 6 (38) | 6 (32) | 22 (132)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 4 (21) | 6 (23) | 6 (23) | 16 (75)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 2 (2) | 8 (12)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (10) | 5 (13) | 4 (12) | 11 (34)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 3 (5) | 3 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 7 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (7) | 5 (12) | 4 (4) | 12 (21)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (5) | 5 (12) | 1 (1) | 12 (30)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (7) | 1 (1) | 1 (1) | 8 (15)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (11) | 3 (6) | 4 (7) | 19 (46)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 3 (3) | 7 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (10)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 7 (13)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (15)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT02663622/Prot_SAP_000.pdf